CLINICAL TRIAL: NCT03546010
Title: Oculometry as an Attentional Mechanism Evaluation Tool and Attention Deficit Hyperactivity Inhibition
Acronym: TDAH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 38RC14.100
Record Dates: First submitted 2018-05-18; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Attention Deficit-Hyperactivity
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oculometric and neuropsychological tests (Experimental): Oculometric tests and neuropsychological tests
  Interventions: Behavioral: Neuropsychological tests; Behavioral: Oculometric tests

INTERVENTIONS:
Behavioral: Neuropsychological tests — WISC test, BRIEF test, NEPSY-2 test, TAP2.3 test, Teach test
Behavioral: Oculometric tests — When the subject see a peripheric target, he should take a look not at the target but in the controlateral half-field, at a mirror position. This is called an anti-saccade task.

SUMMARY:
The aim of this study is to analyse thanks to eye tracking experiments ocular movement classical parameters in children with attention deficit hyperactivity (ADH) and to compare them to results obtained in healthy children and to results obtained with neuropsychological tests commonly used in standard health care.

We should then be able to compare eye tracking with neuropsychological parameters.

The final objective is to give to health professional a tool for ADH investigation with which they should be able to do a simple and effective follow up of children with ADH.

ELIGIBILITY:
Inclusion Criteria:

* Children between 8 and 12 years old
* Boys and girls
* DSM-IV-TR diagnostic criteria for ADH
* Children with methylprednisone treatment
* Social security affiliation
* signed informed consent

Exclusion Criteria:

* specialised scholarship
* refusal from children or parents
* too law results in WISC test (pre-inclusion test)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2014-05-05 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between oculometric and neuropsychological tests in ADH evaluation | Day 1
  Differentiation between simple oculomotor disorder and attentional-visual disorder

CONTACTS AND LOCATIONS:
Overall Officials: Annie Laurent, MD, Principal Investigator — Grenoble Alps University Hospital
Locations (1):
- Grenoble Alps Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malsert J, Guyader N, Chauvin A, Polosan M, Szekely D, Bougerol T, Marendaz C. Saccadic performance and cortical excitability as trait-markers and state-markers in rapid cycling bipolar disorder: a two-case follow-up study. Front Psychiatry. 2013 Jan 4;3:112. doi: 10.3389/fpsyt.2012.00112. eCollection 2012. PMID 23293609